CLINICAL TRIAL: NCT04539769
Title: Impact of the Type of Reconstruction Methods on Diabetes Following Laparoscopic Distal Gastrectomy in Patients With Gastric Cancer and Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyungpook National University Chilgok Hospital (Other)
Collaborators: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Ji Yeon Park, Dr., Kyungpook National University Chilgok Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNUCH 2017-07-011
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Stomach Neoplasms; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Stomach Neoplasms; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BI group (Active Comparator): Conventional Billroth I reconstruction
  Interventions: Procedure: conventional BI
- BII group (Experimental): Billroth II reconstruction with 100-cm long biliopancreatic limb
  Interventions: Procedure: long-limb BII
- RY group (Experimental): Roux-en-Y reconstruction with 100-cm long Roux limb
  Interventions: Procedure: long-limb RY group

INTERVENTIONS:
Procedure: conventional BI — After standard laparoscopic distal gastrectomy with radical lymphadenectomy, the gastrointestinal continuity will be restored with conventional Billroth I gastroduodenostomy.
  Arms: BI group
Procedure: long-limb BII — After standard laparoscopic distal gastrectomy with radical lymphadenectomy, the gastrointestinal continuity will be restored with Billroth II gastrojejunostomy using 100 cm-long biliopancreatic limb.
  Arms: BII group
Procedure: long-limb RY group — After standard laparoscopic distal gastrectomy with radical lymphadenectomy, the gastrointestinal continuity will be restored with Roux-en-Y reconstruction using 100 cm-long Roux limb and standard biliopancreatic limb.
  Arms: RY group

SUMMARY:
There is a rapidly growing interest in metabolic surgery for the treatment of type 2 diabetes. However, its efficacy in the non-morbidly population is not clear yet and the underlying mechanism remains elusive.

Meanwhile, the incidence of early gastric cancer (EGC) in Korea has gradually increased, the long-term quality of life of the patients with EGC has become an important issue. Since the reconstruction methods after gastric cancer surgery are similar to that of metabolic surgery, some surgeons have attempted to modify the reconstruction methods after standard radical gastrectomy to achieve better glycemic control in gastric cancer patients with type 2 diabetes.

The present study aimed to investigate the changes in glucose metabolism and incretin hormone responses following different types of reconstruction after distal gastrectomy in non-morbidly obese gastric cancer patients with type 2 diabetes. This is a non-randomized, prospective, single-center, phase II pilot study.

Patients diagnosed with stage I gastric cancer and type 2 diabetes are eligible for the present study. Patients who will undergo laparoscopic distal gastrectomy for cancer located at the lower two-thirds of the stomach will only be included. The reconstruction method will be selected among conventional Billroth I, long-limb Billroth II (with 100 cm-long biliopancreatic limb), or long-limb Roux-en-Y (with 100 cm-long Roux limb) reconstruction methods according to the surgeon's preference as well as the size of the remnant stomach. All the patients are subjected to a 75g-oral glucose tolerance test (OGTT) preoperatively, and at 5 days, 3 months, 6 months postoperatively and serum glucose, as well as incretin hormones, will be serially measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes as well as pathologically proven gastric cancer of clinical stage I according to the AJCC 7th edition
* Those who are expected to undergo laparoscopic distal gastrectomy
* Body mass index < 30 kg/m2

Exclusion Criteria:

1. baseline fasting C-peptide level < 1.0 ng/dL (who had the possibility of type 1 diabetes)
2. previous radiotherapy or surgery at upper abdomen other than laparoscopic cholecystectomy
3. other malignancies in recent 5 years
4. vulnerable patients (pregnant women, those with cognitive impairment, etc)
5. ECOG-PS ≥ 2
6. participating in other clinical trials within 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Diabetes remission rate | at 6 months after surgery
  the rate of patients achieving HbA1c < 6.5% without antidiabetic medications

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Chilgok Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided